CLINICAL TRIAL: NCT07355270
Title: A U.S. Pilot Human Investigation of RadiofrEquency Vapor Ablation System to Evaluate Safety, TOleRability, and Effectiveness for Proximal Intestinal Mucosal Ablation in Patients With Type 2 Diabetes Mellitus (RESTORE-1 Study)
Acronym: RESTORE-1
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aqua Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLD-1021-US
Record Dates: First submitted 2026-01-20; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Type-2 Diabetes Mellitus
Keywords: RESTORE-1; Type-2 Diabetes Mellitus; T2DM; Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Open label, prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Study arm- RF Vapor Ablation arm (PIMA arm) (Experimental): This is a single arm study. All enrolled patients will be included in this arm
  Interventions: Device: RF Vapor Ablation

INTERVENTIONS:
Device: RF Vapor Ablation — RF Vapor ablation of the proximal intestinal mucosa
  Other Names: Aqua Medical RF Vapor System

SUMMARY:
The purpose of this study is to assess the safety, tolerability and effectiveness of RF vapor ablation of the proximal intestinal mucosa. This study will test the hypothesis that RF vapor ablation will result in improvement in glycemic parameters, without Serious Adverse Events (SAE) or Unanticipated Adverse Device Effects (UADE).

DETAILED DESCRIPTION:
The main aims of the study are :

Evaluate the safety of the device and procedure based on the reported adverse events that occur.

Evaluate device tolerability based on pain scores reported by patients. Evaluate the effectiveness of the device and procedure by comparing change in HbA1c from baseline to 168 days post procedure.

The subject population for this study are adults (22-65 years of age) with type-2 diabetes mellitus. Study participation is 6 months for each patient.

The study is comprised of 5 phases: Screening, Run-in, Pre-procedure tests, RF Vapor ablation procedure, and Post-vapor ablation follow-up (up to 168 days).

ELIGIBILITY:
Inclusion Criteria:

1. Men and non-pregnant women 22-65 years of age
2. Diagnosed with T2DM for at least 1 year and less than or equal to 15 years
3. HbA1C of 7.5 - 10% (58-86 mmol/mol)
4. BMI ≥ 24 and ≤ 40 kg/m2
5. On one or more non-insulin glucose-lowering medications, with no therapeutic changes in medication regimen for at least 12 weeks prior to the screening visit, to ensure stable glycemic control.

   Note 1: Exception for sulfonylureas (SU): For safety reasons, subjects taking sulfonylureas (limited to glipizide or glimepiride only) will be required to undergo a protocol-mandated reduction to ≤50% of the maximum labeled dose during the run-in phase. This adjustment is intended solely to minimize the risk of hypoglycemia during intensive monitoring and dietary standardization and will not be considered a therapeutic change for purposes of eligibility. Subjects unwilling to comply with this dose reduction will be excluded.

   Note 2: GLP-1s are considered non-insulin glucose lowering medications.
6. Agrees to use an additional glucose-lowering treatment (e.g., liraglutide, other OAD except for glyburide), if recommended by the study Investigator in case of persistent hyperglycemia.
7. Weight stability (defined as a < 5% change in body weight) in the 12 weeks prior to the screening visit. Participants should agree to refrain from using over the counter or herbal supplements intended for weight loss. Participants already on a prescribed weight loss drug should agree to not further titrate their medications during the study.
8. Women of childbearing potential must be using at least one acceptable method of contraception throughout the study
9. Willing and able to use CGM for the duration of the study and comply with study visits and study tasks as required per protocol.
10. Able to comply with study requirements and understand and sign the Informed Consent Form

Exclusion Criteria:

1. Diagnosis of Type-1 Diabetes
2. History of diabetic ketoacidosis or hyperosmolar nonketotic coma.
3. Probable insulin production failure, defined as serum C-peptide of 0.3-0.6 nmol/l.
4. Current or previous use of any types of insulin for >1 month (at any time, except for treatment of gestational diabetes) in the last 2 years.
5. Hypoglycemia unawareness as defined by a score of 4 or higher on a Gold score questionnaire suggestive of impaired awareness of hypoglycemia (IAH).
6. History of severe hypoglycemia (2 or more severe hypoglycemic event, as defined by need for third-party assistance, in the last 6 months from the screening visit).
7. Subjects with untreated or unstable microvascular complications of diabetes such as retinopathy, nephropathy, and neuropathy. Subjects who have been appropriately treated/monitored and stable for the prior 3 months before study participation can be included as determined as safe and reasonable by the study PI.
8. Known systemic autoimmune disease that is uncontrolled or requiring steroids or biologics, including a positive anti-glutamic acid decarboxylase (GAD) test. Systemic autoimmune diseases include but not limited to celiac disease, duodenal Crohn disease or pre-existing symptoms of systemic lupus erythematosus, scleroderma or other systemic autoimmune connective tissue disorder. (Participants with adequately controlled primary hypothyroidism or with mild to moderate psoriasis managed with topical therapy-affecting less than 10% of body surface area and not involving special areas (e.g., face, palms)-may be included).
9. Previous GI surgery that could limit access to the duodenum such as Billroth 2, Roux-en-Y gastric bypass, or other similar procedures or conditions. (Patients who have undergone a laparoscopic sleeve gastrectomy (LSG) or an endoscopic sleeve gastrectomy (ESG) procedure more than one year prior to enrollment will not be excluded from participation in this study.)
10. History of chronic pancreatitis or a diagnosis of idiopathic acute pancreatitis within the past 12 months.
11. Documented history of diabetic gastroparesis confirmed by gastric emptying study.
12. Known active hepatitis or liver disease, excluding nonalcoholic steatohepatitis (NASH) and nonalcoholic fatty liver disease (NAFLD).
13. Symptomatic gallstones, or acute gastrointestinal illness in the previous 7 days.
14. Known history of severe irritable bowel syndrome, radiation enteritis or other inflammatory bowel syndrome, such as Crohn's disease and Celiac disease.
15. Alcoholic liver disease, as indicated by ANI>-0.66 and AUDIT-C questionnaire
16. Known history of a structural or functional esophageal disorder that could impede endoscope passage or elevate the risk of esophageal injury during an endoscopic procedure, including but not limited to moderate-severe (Los Angeles Grade C or D) esophagitis, dysphagia due to achalasia or stricture/stenosis, esophageal varices greater than Grade 2, history of esophageal perforation, or any other clinically significant esophageal condition.
17. Presence of upper gastrointestinal conditions, including active ulcers, varices, strictures, congenital or acquired proximal intestinal telangiectasia, active H. pylori infection.
18. Current use of anticoagulation therapy (vitamin K antagonists, such as warfarin, or current use of direct-action oral anticoagulants (DOACs) that cannot be safely discontinued peri procedurally
19. Current use of P2Y12 inhibitors (clopidogrel, prasugrel, ticagrelor) that cannot be discontinued for 7 days before and 7 days after the procedure.
20. Unable to discontinue high-dose non-steroidal anti-inflammatory drugs (NSAIDs) during treatment through 4 weeks following the procedure. Use of acetaminophen and low dose aspirin, PRN over the counter NSAIDs is allowed.
21. Use of systemic glucocorticoids (excluding topical or ophthalmic application or inhaled forms) for more than 10 consecutive days within 12 weeks prior to the baseline visit.
22. Persistent anemia, defined as hemoglobin <10 g/dl on two consecutive measurements >6 weeks apart.
23. Known history of hemoglobinopathy.
24. Known history of blood donation or transfusion within 3 months prior or screening or anticipated blood donation during the study period.
25. Significant cardiovascular disease, including known history of valvular heart disease, or myocardial infarction, heart failure, transient ischemic attack, or stroke within 12 months prior to the Screening Visit.
26. Mean of 3 separate blood pressure measurements >180 mmHg (systolic) or >100 mmHg (diastolic).
27. Estimated glomerular filtration rate (eGFR) ≤ 45 ml/min/1.73m2 (estimated by MDRD).
28. Known immunocompromised status, including but not limited to: individuals who have undergone organ transplantation, receipt of chemotherapy, or radiotherapy within the past 12 months, clinically significant leukopenia, confirmed human immunodeficiency virus (HIV) infection, or any other condition impacting immune function that, in the opinion of the investigator, renders the participant unsuitable for trial participation.
29. History of secondary hypothyroidism or inadequately controlled primary hypothyroidism (TSH value >1.5x of the upper limit of normal range at screening)
30. In the opinion of the Investigator, the participant is not an appropriate candidate for upper GI endoscopy or general anesthesia.
31. Active illicit substance abuse or Alcohol Use Disorder (AUD) (consuming more than 14 drinks per week for men or more than seven drinks per week for women)
32. Active malignancy within the last 5 years (excluding non-melanoma skin cancers)
33. Women who are currently breastfeeding
34. Participating in another ongoing clinical trial of an investigational drug or device.
35. Any other physical or mental condition that, in the opinion of the investigator, would make the participant an unsuitable candidate for clinical trial participation.
36. Critically ill or has a life expectancy <3 years.
37. Use of a cardiac pacemaker, implantable cardioverter-defibrillator (AICD), duodenal metallic implants, or any other implanted electronic medical devices.
38. General contraindications to deep or conscious sedation, general anesthesia, or upper gastrointestinal (GI) endoscopy, including individuals deemed high-risk by an anesthesiologist (e.g., ASA Physical Status Classification of IV or higher).

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Safety endpoint | 6 months
  Number of subjects with reported device or procedure related SAEs or UADEs.
Tolerability endpoint | 14 days
  Descriptive statistics on Visual Analogue Scale(VAS) pain scores (A Visual Analog Scale (VAS) pain score is a patient's self-reported measure of pain intensity, marked on a straight line scale from 0-10, with "no pain" at the zero-end and "worst imaginable pain" at 10.)
Efficacy endpoint | 6 months
  Change in HbA1c from baseline to 6 months post procedure

SECONDARY OUTCOMES:
Change in HbA1c at 3 months post procedure | 3 months
  Change in HbA1c (from baseline) at 3 months post procedure will be analyzed
Change in FPG from baseline to 3 months and 6 months post procedure | 6 months
  Change in Fasting Plasma Glucose from baseline to 3 months and 6 months post procedure
Proportion of ablation-treated subjects with an HbA1c improvement > 0.5% from baseline at 6 months. | 6 months
  Proportion of ablation-treated subjects with an HbA1c improvement > 0.5% from baseline at 6 months.
Change in HOMA-IR from baseline to 6 months post procedure. | 6 months
  Change in HOMA-IR from baseline to 6 months post procedure.
Change in UACR from baseline to 6 months post procedure. | 6 months
  Change in Urine Albumin-Creatinine Ratio from baseline to 6 months post procedure.
Change in ALT and AST from baseline to 6 months post procedure. | 6 months
  Change in ALT and AST from baseline to 6 months post procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Shaheen, MD, Principal Investigator — University of North Carolina
Locations (2):
- United States (2):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - University of North Carolina School of Medicine, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers.